CLINICAL TRIAL: NCT05036694
Title: Diagnostic Performance of a Novel Lipoarabinomannan Test (FujiLAM) to Detect Tuberculosis in HIV-positive Patients in Kenya
Brief Title: Diagnostic Performance of a Novel Lipoarabinomannan.
Acronym: FUJILAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Médecins Sans Frontières, Kenya (Other)
Collaborators: Epicentre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANRS12429
Record Dates: First submitted 2021-07-08; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-07

CONDITIONS: HIV Primary Infection
Keywords: TUBERCULOSIS IN HIV

STUDY DESIGN:
Intervention Model Description: GROUP 1_ TB SYMPTOMS GROUP2_ ADVANCED HIV WITH NO TB SYMPTOMS
Masking Description: We are not blinding the two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulatory HIV positive patients (Other): Ambulatory HIV positive patients with signs and symptoms of TB, and Ambulatory HIV positive patients with advanced disease and CD4 less than 200 cell.
  Interventions: Device: FUJILAM KIT

INTERVENTIONS:
Device: FUJILAM KIT — Urine based test to detect LAM

SUMMARY:
The Fujifilm SILVAMP TB LAM (FujiLAM; Fujifilm, Tokyo, Japan) is a novel (not commercialized) urine based point-of-care assay to diagnose TB in HIV-positive patients. A first study using urine frozen samples has reported a higher sensitivity of this test over the currently commercialised Alere Determine TB LAM Ag assay (AlereLAM).

DETAILED DESCRIPTION:
The study aims to assess the performance of a new test called the Fujifilm SILVAMP TB LAM or simply the Fuji-LAM test. The Fuji-LAM test is a test that can be done on urine to look for specific proteins that are produced by the bacteria that causes tuberculosis. This test offers an advantage over the tests that are based on phlegm because most patients can produce urine for testing even when they are very sick. Additionally, this test does not require a complex laboratory set up and it can therefore be used by health workers as they interact with the patient. This study will also look at how the new test compares with an existing test AlereLAM - that is based on similar technology. Initial laboratory-based studies conducted on frozen urine samples show that the new test has better performance than the existing test. This study is different from the first studies because it is being conducted in real life settings rather than in a laboratory.

The study will be conducted at the Homa Bay County Hospital in Kenya. Individuals living with HIV with and without signs and symptoms of TB will be invited to take part. Individuals who agree to participate will be seen by the health workers in the study and will provide samples for testing using the FujiLAM test and other standard tests used to investigate individuals for suspected tuberculosis.

Investigators are also conducting similar studies in other African countries including Uganda, Mozambique and South Africa. This will enable investigators to assess the performance of the test in diverse settings.

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age or older
* HIV-positive Group 1: At least one symptom of TB

Group 2:

* Advanced HIV disease (CD4 count less than 200cell/µl or clinical stage III/IV)
* No signs and symptoms of TB
* Signature of the informed consent

Exclusion Criteria:

* Intake of anti-tuberculosis drugs for more than 5 days in the month prior to the consultation except preventive TB treatment.
* Decline to sign informed consent.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the diagnostic performance of FujiLAM in ambulatory HIV positive patients. | 12 months
  Proportion of patients with a positive FujiLAM result among patients with microbiologically confirmed TB in ambulatory HIV-positive patients with signs and symptoms of TB (Group 1) and Diagnostic performance of FujiLAM test to detect tuberculosis in HIV-positive patients in Kenya - Protocol v2.3 14 in ambulatory HIV-positive patients with advanced HIV disease and no signs and symptoms of TB (Group 2).

SECONDARY OUTCOMES:
To assess the sensitivity of FujiLAM at different levels of CD4 count. | 12 months
  * Proportion of patients with a positive FujiLAM result among patients with probable TB or microbiologically confirmed TB in ambulatory HIV-positive patients with signs and symptoms of TB (Group 1) and in ambulatory HIV-positive patients with advanced HIV disease and no signs and symptoms of TB (Group 2).
  * Proportion of patients with a positive FujiLAM result among patients with microbiologically confirmed TB and among patients with probable TB or microbiologically confirmed TB by level CD4.
  * Proportion of patients with a positive AlereLAM among patients with microbiologically confirmed
  * TB and among patients with probable TB or microbiologically confirmed TB by level of CD4.

CONTACTS AND LOCATIONS:
Overall Officials: HELENA DR Coordinating Principal Investigator, PhD, Principal Investigator — MEDECIN SAN FRONTIERES